CLINICAL TRIAL: NCT00430807
Title: Multicentric Double Blind Versus Placebo Randomised Study Evaluating the Corticosteroid Sparing Effect of Hydrocyschloroquine in Non Complicated Giant Cell Arteritis.
Brief Title: Hydroxychloroquine in Giant Cell Arteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0102808; PHRC 2001 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Giant Cell Arteritis
Keywords: giant cell arteritis,; hydroxychloroquine,; corticosteroid sparing,; corticodependence
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydroxychloroquine/placebo

SUMMARY:
Cortico-dependence is frequent in giant cell arteritis patients, and no drugs has proved its ability to prevent corticodependence. Hydrocychloroquine is a well tolerated immunomodulatory drug that may have a corticosteroid sparing potential according to immuno-pharmacological and clinical data. We have designed a multcentric double blind versus placebo randomized controled trial to assess the corticosteroid sparing effect of hydroxychloroquine in non complicated giant cell arteritis.

ELIGIBILITY:
Inclusion Criteria:

* giant celle arteritis with at least 3 ACR criteria including a disgnostic temporal artery biopsy
* corticosteroid treatment since less than 1 month
* age less than 85 years
* signed informed consent

Exclusion Criteria:

* amaurosis fugax, loss of vision, acute lumb ischemia, angina pectoris or myocardium infarctus, mesenteric ischemia or other vascular complications related to GCA
* low life expectancy (<2 years)
* corticosteroid treatment since more than 30 days whatever the dosage
* primary corticosteroid resistance defined by persistant symptoms despite prednisone for more than 15 days
* previous psychiatric troubles induced corticosteroids
* hydroxychloroquine contra-indicated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-01; Primary Completion 2005-01 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
prednisone dosage equal to or lower than 5 mg since more than 3 months without | 3 months at least
having experienced relapse since the inclusion in the study

SECONDARY OUTCOMES:
prednisone daily dosage | 6, 12, 18 and 24 months
hydroxychloroquine blood levels

CONTACTS AND LOCATIONS:
Overall Officials: ARLET Philippe, D, Principal Investigator — CHU Toulouse, Hôpital Purpan; SAILLER Laurent, MD, Study Director — CHU Toulouse, Service de Médecine Interne, Hôpital Purpan
Locations (23):
- France (23):
  - Hospital, Agen
  - Hospital, Albi
  - Hospital Auch, Auch
  - Hospital Avignon, Avignon
  - University Hospital Besançon, Besançon
  - Hospital Béziers, Béziers
  - University Hospital Côte de Nacre, Caen
  - University Hospital Dijon, Dijon
  - Hospital, Foix
  - Hospital, Lavaur
  - University Hospital Dupuytren, Limoges
  - Hospital, Lisieux
  - Hospital, Lourdes
  - Hospital, Mazamet
  - Hospital, Montauban
  - University Hospital, Nantes
  - Saint Louis Hospital, Paris
  - University Hospital Saint Antoine, Paris
  - University Hospital Bichat, Paris
  - Hospital Suresnes, Suresnes
  - University Hospital Toulouse, Toulouse
  - University Hospital, Toulouse
  - University Hospital Bretonneau, Tours

REFERENCES:
- [Background] Jover JA, Hernandez-Garcia C, Morado IC, Vargas E, Banares A, Fernandez-Gutierrez B. Combined treatment of giant-cell arteritis with methotrexate and prednisone. a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2001 Jan 16;134(2):106-14. doi: 10.7326/0003-4819-134-2-200101160-00010. PMID 11177313
- [Background] Chevalet P, Barrier JH, Pottier P, Magadur-Joly G, Pottier MA, Hamidou M, Planchon B, El Kouri D, Connan L, Dupond JL, De Wazieres B, Dien G, Duhamel E, Grosbois B, Jego P, Le Strat A, Capdeville J, Letellier P, Agron L. A randomized, multicenter, controlled trial using intravenous pulses of methylprednisolone in the initial treatment of simple forms of giant cell arteritis: a one year followup study of 164 patients. J Rheumatol. 2000 Jun;27(6):1484-91. PMID 10852275
- [Background] Mazlumzadeh M, Hunder GG, Easley KA, Calamia KT, Matteson EL, Griffing WL, Younge BR, Weyand CM, Goronzy JJ. Treatment of giant cell arteritis using induction therapy with high-dose glucocorticoids: a double-blind, placebo-controlled, randomized prospective clinical trial. Arthritis Rheum. 2006 Oct;54(10):3310-8. doi: 10.1002/art.22163. PMID 17009270
- [Background] Le Guennec P, Dromer C, Sixou L, Marc V, Coustals P, Fournie B. [Treatment of Horton disease. Value of synthetic antimalarials. Apropos of a retrospective study of 36 patients]. Rev Rhum Ed Fr. 1994;61(7-8):485-90. French. PMID 7833883
- [Background] David-Chausse J, Dehais J, Leman A. [Results of a regional survey on the treatment of rhizomelic pseudopolyarthritis and temporal arteritis. Apropos of 242 cases treated by various modalities with synthetic antimalarials, corticoids and non-steroidal anti-inflammatory agents]. Rev Rhum Mal Osteoartic. 1983 Jul-Sep;50(8-9):563-71. French. PMID 6635510
- [Background] Hoffman GS, Cid MC, Hellmann DB, Guillevin L, Stone JH, Schousboe J, Cohen P, Calabrese LH, Dickler H, Merkel PA, Fortin P, Flynn JA, Locker GA, Easley KA, Schned E, Hunder GG, Sneller MC, Tuggle C, Swanson H, Hernandez-Rodriguez J, Lopez-Soto A, Bork D, Hoffman DB, Kalunian K, Klashman D, Wilke WS, Scheetz RJ, Mandell BF, Fessler BJ, Kosmorsky G, Prayson R, Luqmani RA, Nuki G, McRorie E, Sherrer Y, Baca S, Walsh B, Ferland D, Soubrier M, Choi HK, Gross W, Segal AM, Ludivico C, Puechal X; International Network for the Study of Systemic Vasculitides. A multicenter, randomized, double-blind, placebo-controlled trial of adjuvant methotrexate treatment for giant cell arteritis. Arthritis Rheum. 2002 May;46(5):1309-18. doi: 10.1002/art.10262. PMID 12115238
- See also: Related Info — http://www.vascularites.org/
- See also: Related Info — http://www.snfmi.org/